CLINICAL TRIAL: NCT05550233
Title: A Prospective, Multicentric, Randomized Controlled Clinical Trial of Drug-coated Balloons in the Treatment of Big de Novo Coronary Artery Disease
Brief Title: Drug-coated Balloons in Big de Novo Coronary Disease
Acronym: DCB-LVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xue Yu, Vice director of cardiology department, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJH-DCB-LVD
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronary Heart Disease
Keywords: drug-coated balloon; de novo coronary disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCB treatment (Experimental): drug-coated balloon in PCI
  Interventions: Device: drug-coated balloon
- DES treatment (Other): drug-eluted stent in PCI
  Interventions: Device: drug-coated balloon

INTERVENTIONS:
Device: drug-coated balloon — drug-coated balloon in big de novo coronary disease
  Other Names: drug-eluted stent

SUMMARY:
A prospective, multicenter, randomized controlled, open-label, non-inferiority trial. Plan to recruit 240 patients whose lesions are de novo coronary artery disease (reference vessel diameter ≥ 3.0 mm), diameter stenosis ≥ 75% with ischemic symptoms or objective evidence of ischemia (ECG, cardionuclide, or FFR), and are suitable for implantation DES or DCB. After successful preconditioning, patients were randomly assigned to two PCI treatment groups(drug-coated balloon or drug-eluted stent) in a 1:1 ratio. The safety and efficacy of drug-coated balloons in PCI treatment of de novo coronary artery lesions (reference diameter 3.0 mm and above) were evaluated by comparing the late lumen loss of two groups of subjects in 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old;
* Asymptomatic myocardial ischemia, stable or unstable angina;
* The subject (or legal guardian) understands the trial requirements and treatment process, and signs a written informed consent before performing any prescribed inspection or operation;
* Willing to undergo all follow-up evaluations requested by the trial, including admission angiographic evaluation at 12 months;
* The target lesion must be the de novo lesion, and the diameter of the reference vessel is ≥3.0mm.

Exclusion Criteria:

* Patients with acute ST-segment elevation myocardial infarction/non-ST-segment elevation myocardial infarction within 3 months;
* Hypersensitivity to the investigational balloon/stent system or concomitant medications required by the protocol;
* Intolerant of dual antiplatelet therapy, or clinical conditions requiring long-term use of oral anticoagulants;
* Life expectancy is less than 12 months;
* eGFR≤30ml/min/1.73m2 or blood purification treatment;
* LVEF≤40% or NYHA cardiac function class≥III;
* Clinical conditions of severe hepatic insufficiency and coagulation disorder
* Pregnant or breastfeeding women;
* Participating in another clinical trial and have not completed the primary endpoint observation of the trial;
* Reference lumen diameter > 4.0mm;
* Branch vessels ≥ 2.0 mm in diameter that may require intervention in the target lesion;
* The vessel where the target lesion is located has an independent lesion with a diameter stenosis of ≥50% and requires interventional therapy;
* Chronic total occlusive disease;
* Left main stem disease;
* Severe calcification, tortuous blood vessels, existing dissection or severe thrombus burden, the investigator judges that DCB is not suitable for treatment of lesions;
* Lesions with failed preprocessing, or lesions whose length exceeds the length of a single DES/DCB need to be covered after preprocessing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
late lumen loss，LLL | 12 months after PCI
  late lumen loss in target lesions obtained by coronary angiography at 12 months after PCI

SECONDARY OUTCOMES:
target lesion failure，TLF | 12 months after PCI
  Cardiac death, target vessel-related myocardial infarction, ischemia-driven target lesion revascularization or target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Fusui Ji, MD, Study Chair — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Published papers